CLINICAL TRIAL: NCT02220309
Title: Neural Dimensions of Threat Reactivity and Regulation for Understanding Anxiety
Brief Title: Stanford RAD-AT Study (Research on Anxiety and Depression - Anhedonia Treatment)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Leanne Williams, Professor, Stanford University
Other Study IDs: 27937
Record Dates: First submitted 2014-08-13; First posted 2014-08-19 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Social Anxiety Disorder; Bipolar disorder II; PTSD; GAD; Phobia
MeSH Terms: conditions — Anxiety Disorders; Depression; Phobia, Social; Bipolar Disorder; Stress Disorders, Post-Traumatic; Phobic Disorders | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — We will collect saliva samples, and in exploratory analysis focus on consideration of genes associated with neuroimaging-behavior constructs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Anxiety and mood disorders
  Interventions: Drug: Pramipexole Oral Tablet

INTERVENTIONS:
Drug: Pramipexole Oral Tablet — Pramipexole is an oral Dopamine agonist.

SUMMARY:
This research study is aimed at understanding behaviors and brain circuits that relate to anxiety and depression. Our goal is to learn which circuits of the brain are involved in anxiety and how these circuits might affect daily functioning.

This study has recently added an additional treatment component: participants undergo a 12 week course of either Pramipexole medication or rTMS therapy (explained below). The ultimate goal of the study is to offer participants experiencing anxiety and depression a treatment that is alternative to ones that have failed them in the past, and to apply the knowledge we gain from investigating the brain circuits involved in anxiety and depression to help personalize treatments.

We invite anyone who has recently experienced any symptoms of anxiety and/or depression to participate (no diagnosis is required to participate).

DETAILED DESCRIPTION:
If you are eligible and choose to participate, we'll ask you to come in for 2 separate testing visits and 8 weeks of treatment in between.

In both the pre-treatment and post-treatment testing visit, you would complete game-like tasks on the computer, undergo a non-invasive MRI brain scan, and answer some questions about your emotional health. The entire visit takes place during 1-2 days at Stanford and lasts about 4-5 hours. We'll also ask you to complete a follow-up 12 weeks later, from home, during which we'll again ask you some questions on your emotional health.

The 8-week treatment phase will consist of your choice of either TMS (transcranial magnetic stimulation) or Pramipexole (a medication for depression). You will meet with study coordinators and MDs each week (Pramipexole) or each day (TMS) to receive treatment. You will also be asked to complete weekly online surveys to monitor your mood during the 2-month course of treatment.

To inquire more about participation, you can either sign up online or contact us.

Sign up online: http://med.stanford.edu/williamslab/research/current/rad.html Contact us: Call or text (650) 600-1609 or email rad-at-study@stanford.edu

ELIGIBILITY:
Inclusion Criteria:

* Recent experiences of anxiety and/or depression
* Ages 18-65

Exclusion Criteria:

* Specific psychiatric medications (case-by-case basis)
* A diagnosis of Bipolar 1 Disorder, Schizophrenia, or Obsessive Compulsive Disorder
* Any of the following medical conditions: Parkinson's disease; liver or kidney disease; history of epilepsy or seizures; history of cardiovascular disorders (specifically orthostatic hypotension)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect to enroll 160 individuals spanning the spectrum of anxiety and associated mood symptoms. These individuals include patients of the Gronowski Center, a community clinical psychology center in Palo Alto. We will also recruit from the community through various advertisements. Further, participants will include healthy people recruited by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2013-08-11; Primary Completion 2024-12-18 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Assessments of symptoms and daily functioning | 12 weeks
  General demographics questionnaires, alcohol use questionnaire, substance use questionnaires, Mood and Anxiety Symptom Questionnaire, Penn State Worry Questionnaire, Health at Work Performance Questionnaire, WHO Quality of Life questionnaire, Satisfaction with Life Survey, Emotion Regulation Questionnaire, Brief COPE questionnaire, Early Life Stress questionnaire, Quick Inventory of Depressive Symptomatology, Beck Depression Inventory, PTSD Checklist - Civilian Version, Beck Anxiety Inventory, Barratt Impulsiveness Scale, MINI Neuropsychiatric Interview
Brain imaging | 12 weeks
  Non-invasive MRI brain scan to see function and structure of brain.
Cognitive assessment | 12 weeks
  WebNeuro is an objective assessment of cognitive strengths and weaknesses. It provides an accurate and objective assessment of person's cognitive function and efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Williams, PhD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Gronowski Center-5150 El Camino Real, Los Altos, California
  - VAPAHCS/Palo Alto MIRECC-3801 Miranda Avenue, Palo Alto, California
  - Stanford University Department of Psychiatry, Stanford, California

REFERENCES:
- [Derived] Williams LM, Goldstein-Piekarski AN, Chowdhry N, Grisanzio KA, Haug NA, Samara Z, Etkin A, O'Hara R, Schatzberg AF, Suppes T, Yesavage J. Developing a clinical translational neuroscience taxonomy for anxiety and mood disorder: protocol for the baseline-follow up Research domain criteria Anxiety and Depression ("RAD") project. BMC Psychiatry. 2016 Mar 15;16:68. doi: 10.1186/s12888-016-0771-3. PMID 26980207
- See also: Research on Anxiety and Depression: The RAD Project — http://williamspanlab.com/rad
- See also: Research on Anxiety and Depression: The RAD Project — http://med.stanford.edu/williamslab/research/current/rad.html